CLINICAL TRIAL: NCT02081378
Title: A Phase I, Multicenter, Open-label Study of Oral ABL001 in Patients With Chronic Myelogenous Leukemia (CML) or Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia (Ph+ ALL)
Brief Title: A Phase I Study of Oral Asciminib (ABL001) in Patients With CML or Ph+ ALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001X2101; 2013-004491-36 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-07 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Myelogenous Leukemia; Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Keywords: CML; Ph+ ALL; asciminib; ABL001; Maximum Tolerated Dose (MTD); Recommended Dose for Expansion (RDE); relapsed or refractory; TKIs; Nilotinib; Imatinib; Dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Recurrence | interventions — asciminib; nilotinib; Imatinib Mesylate; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Asciminib in CML patients (Experimental): Dose escalation study estimated the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of asciminib in adult patients with chronic myeloid leukemia (CML).
  Interventions: Drug: Asciminib (ABL001)
- Asciminib+Nilotinib in CML patients (Experimental): Dose escalation study estimated the MTD and/or RDE of asciminib in combination with Nilotinib in adult CML patients
  Interventions: Drug: Asciminib (ABL001); Drug: Nilotinib
- Asciminib in Ph+ ALL patients (Experimental): Dose escalation study estimated the MTD and/or RDE of asciminib in adult patients with Ph positive ALL patients
  Interventions: Drug: Asciminib (ABL001)
- Asciminib+Imatinib in CML patients (Experimental): Dose escalation study to estimate the MTD and/or RDE of asciminib in combination with imatinib in adult CML patients
  Interventions: Drug: Asciminib (ABL001); Drug: Imatinib
- Asciminib+dasatinib in CML patients (Experimental): Dose escalation study estimated the MTD and/or RDE of asciminib in combination with dasatinib in adult CML patients
  Interventions: Drug: Asciminib (ABL001); Drug: Dasatinib

INTERVENTIONS:
Drug: Asciminib (ABL001) — Asciminib was be administered orally in a dose escalation schedule.
  Other Names: ABL001
Drug: Nilotinib — Asciminib and Nilotinib was administered orally in CML patients
  Arms: Asciminib+Nilotinib in CML patients
Drug: Imatinib — Asciminib and imatinib was administered orally in CML patients
  Arms: Asciminib+Imatinib in CML patients
Drug: Dasatinib — Asciminib and dasatinib was administered orally in CML patients
  Arms: Asciminib+dasatinib in CML patients

SUMMARY:
The design of a phase I, open label, dose finding study was chosen in order to establish a safe and tolerated dose of single agent ABL001 in Chronic myeloid leukemia (CML) and Philadelphia chromosome positive Acute lymphoblastic leukemia (Ph+ ALL) patients who are relapsed or refractory to or are intolerant of Tyrosine kinase inhibitors (TKIs), and of ABL001+Nilotinib, ABL001+Imatinib and ABL001+Dasatinib in Ph positive CML patients who are relapsed or refractory to TKIs.

DETAILED DESCRIPTION:
This first-in-human trial with ABL001 was a dose escalation study whose primary purpose was to estimate the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of single agent ABL001 in CML or Ph+ ALL patients, and in combination with either Nilotinib or Imatinib or Dasatinib in Ph positive CML patients. The safety, tolerability and pharmacokinetic (PK) profile of ABL001 and ABL001+Nilotinib, ABL001+Imatinib and ABL001+Dasatinib were assessed together with an evaluation of pharmacodynamic (PD) changes in peripheral blood mononuclear cells (PBMC) and bone marrow aspirates and all data could contribute to the assessment of the RDE.

An understanding of the MTD/RDE, safety profile, PK/PD relationship, and preliminary evidence of anti-CML and ALL activity wias used to inform future development in adults with CML and Ph+ ALL. By virtue of its distinct pharmacological profile and by preclinical pharmacological studies demonstrating an additive effect, a combination of ABL001 and a tyrosine-kinase inhibitor (TKI) has the potential to achieve a deeper molecular response in a higher proportion of CML patients as compared to single agent TKI therapy. Such a combination has the added advantage of targeting the ABL kinase domain at two distinct locations, theoretically preventing single point mutation-associated treatment resistance. The prediction is that a nilotinib+ABL001, imatinib+ABL001 and/or dasatinib+ABL001 combination will increase the percentage of patients who achieve a complete molecular response (CMR) and decrease the time to CMR, thereby increasing the possibility of achieving sustained treatment-free remissions in these patients. In addition, some patients could be intolerant of therapy with TKIs or could develop mutations that promote resistance to TKI therapy. In these patients, ABL001 could provide a novel therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

For CML patients either:

* a. Patients with Ph+ CML in chronic or accelerated phase who were previously treated with at least two different tyrosine kinase inhibitors prior to study entry and are relapsed, refractory to or intolerant of TKIs as determined by investigators or
* b. Patients with CML in chronic or accelerated phase who exhibit relapsed disease associated with the presence of the T315I "gatekeeper mutation" after at least one TKI are also eligible provided that no other effective therapy exists

For ALL and CML-BP patients:

* Patients with CML BP or Ph+ ALL who have a cytopathologically confirmed diagnosis and are relapsed or refractory to at least one prior TKI or intolerant of TKIs. TKI failure for Ph+ ALL and CML-BP patients is defined as at least the loss of Molecular Response (MR) 4.5 (BCR-ABL ≤ 0.0032%)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Willingness and ability to comply with all study procedures
* Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

Wash-out period:

* Systemic antineoplastic therapy (including cytotoxic chemotherapy, alfa-interferon and toxin immunoconjugates) or any experimental therapy within 14 days or 5 half-lives, whichever is shorter, before the first dose of study treatment
* Therapy with TKIs as single agent within 5 half-lives before the first dose of study treatment
* Unconjugated monoclonal antibody therapies within 28 days or 5 half-lives, whichever is shorter, before the first dose of study treatment
* For patients receiving ABL001 in combination with either nilotinib or imatinib or dasatinib, intolerance to nilotinib, imatinib or dasatinib, respectively
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment.
* CNS irradiation for meningeal leukemia, except if radiotherapy occurred > 3 months previously. At least four weeks must have elapsed since prophylactic CNS irradiation given as part of a front-line therapy regimen for ALL
* Major surgery within 2 weeks before the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) during the first cycle of study treatment | First Cycle is 28 days
  Determine the MTD and/or RDE of ABL001 as single agent in CML and Ph+ ALL, and in combination with either nilotinib or imatinib or dasatinib in CML patients

SECONDARY OUTCOMES:
Hematologic Response | At screening and first day of cycle 2 and 3 and every 12 weeks afterwards
Cytogenetic response | at screening or when a patient's BCR-ABL ratio has risen to >1%
BCR-ABL transcript level | At screening and first day of cycle 2 and 3 and every 12 weeks afterwards
Cmax of ABL001 as measured in plasma | Cycle 1 days 1,2,8,15,16 and 22. Cycle 2 days 1 and 2, and subsequent cycles at the begining of each cycle up to cycle 6.
Cmin of ABL001 as measured in plasma | Cycle 1 days 1,2,8,15,16 and 22. Cycle 2 days 1 and 2, and subsequent cycles at the begining of each cycle up to cycle 6.
AUCinf of ABL001 as measured in plasma | Cycle 1 days 1,2,8,15,16 and 22. Cycle 2 days 1 and 2, and subsequent cycles at the begining of each cycle up to cycle 6.
AUClast of ABL001 as measured in plasma | Cycle 1 days 1,2,8,15,16 and 22. Cycle 2 days 1 and 2, and subsequent cycles at the begining of each cycle up to cycle 6.
AUCtau of ABL001 as measured in plasma | Cycle 1 days 1,2,8,15,16 and 22. Cycle 2 days 1 and 2, and subsequent cycles at the begining of each cycle up to cycle 6.
T1/2 of ABL001 as measured in plasma | Cycle 1 days 1,2,8,15,16 and 22. Cycle 2 days 1 and 2, and subsequent cycles at the begining of each cycle up to cycle 6.
Adverse events | Collected from screening visit through post-treatment follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (6):
  - Dana Farber Cancer Institute Hematology / Oncology, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center SC, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center Memorial Sloan Kettering, New York, New York
  - Oregon Health Sciences University SC-6, Portland, Oregon
  - University of Texas/MD Anderson Cancer Center UT MD Anderson, Houston, Texas
  - Huntsman Cancer Institute SC, Salt Lake City, Utah
- Novartis Investigative Site, Adelaide, South Australia, Australia
- France (2):
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Bordeaux
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Jena
- Novartis Investigative Site, Roma, RM, Italy
- Novartis Investigative Site, Kobe, Hyōgo, Japan
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Seocho Gu, South Korea
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luskin MR, Murakami MA, Keating J, Flamand Y, Winer ES, Garcia JS, Stahl M, Stone RM, Wadleigh M, Jaeckle SL, Hagopian E, Weinstock DM, Liegel J, McMasters M, Wang ES, Stock W, DeAngelo DJ. Asciminib plus dasatinib and prednisone for Philadelphia chromosome-positive acute leukemia. Blood. 2025 Feb 6;145(6):577-589. doi: 10.1182/blood.2024025800. PMID 39374521
- [Derived] Li YF, Combes FP, Hoch M, Lorenzo S, Sy SKB, Ho YY. Population Pharmacokinetics of Asciminib in Tyrosine Kinase Inhibitor-Treated Patients with Philadelphia Chromosome-Positive Chronic Myeloid Leukemia in Chronic and Acute Phases. Clin Pharmacokinet. 2022 Oct;61(10):1393-1403. doi: 10.1007/s40262-022-01148-9. Epub 2022 Jun 28. PMID 35764773
- [Derived] Hughes TP, Mauro MJ, Cortes JE, Minami H, Rea D, DeAngelo DJ, Breccia M, Goh YT, Talpaz M, Hochhaus A, le Coutre P, Ottmann O, Heinrich MC, Steegmann JL, Deininger MWN, Janssen JJWM, Mahon FX, Minami Y, Yeung D, Ross DM, Tallman MS, Park JH, Druker BJ, Hynds D, Duan Y, Meille C, Hourcade-Potelleret F, Vanasse KG, Lang F, Kim DW. Asciminib in Chronic Myeloid Leukemia after ABL Kinase Inhibitor Failure. N Engl J Med. 2019 Dec 12;381(24):2315-2326. doi: 10.1056/NEJMoa1902328. PMID 31826340
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18152